CLINICAL TRIAL: NCT02438501
Title: A Prospective, Randomized, Open-label, Multi-center Study of Efficacy of Palliative Low-Dose Involved-Field Radiation Therapy for Recurrent Advanced Follicular Lymphoma: Wuhan University Cancer Center -NHL02 Trial
Brief Title: Efficacy of Palliative Low-Dose Involved-Field Radiation Therapy for Recurrent Advanced Follicular Lymphoma
Acronym: WUCC-NHL02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Di Deng (Other)
Responsible Party: Sponsor-Investigator, Di Deng, Associate Professor, Director of Research, Wuhan University
Organization: Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WuhanU
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Recurrent Follicular Lymphoma
Keywords: low-dose involved field radiotherapy; recurrent; advanced; follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LD-IFRT group (Experimental): Chemotherapy / Low-dose involved-field radiotherapy
  Interventions: Radiation: Low-dose involved-field radiotherapy
- IFRT group (Active Comparator): Chemotherapy / Involved-field radiotherapy
  Interventions: Radiation: Involved-field radiotherapy

INTERVENTIONS:
Radiation: Low-dose involved-field radiotherapy — Low-dose involved-field RT (LD-IFRT) is given in 2 daily fractions (2×2 Gy). Involved-field of radiotherapy defined by CALGB is encompassed the prechemotherapy gross tumor.
  Arms: LD-IFRT group
Radiation: Involved-field radiotherapy — Involved-field RT (IFRT) is given in 24 Gy in 12 fractions. Radiotherapy field defined by CALGB is encompassed the prechemotherapy gross tumor.
  Arms: IFRT group

SUMMARY:
Many trials that patients with advanced or recurrent indolent lymphoma managed with very low-dose (4Gy) limited-field RT (LD-IFRT) have shown that high response rates and durable remission can be achieved. However, the results of two phase III trials have failed to demonstrate the lasting response rate (RR) with LD-IFRT versus in other approaches. Histology, bulky tumor (>5 cm), higher number of prior chemotherapy regimens, adoption of rituximab, and age>65 years have been shown to significantly influence response rates of LD-IFRT. The objectives of this trial investigate the efficacy of palliative low-dose involved-field radiation therapy in patients lower than 65 years of age with recurrent advanced follicular lymphoma.

DETAILED DESCRIPTION:
Introduction: Follicular lymphoma（FL) often involves lymph nodes and the bone marrow and is widely regarded as a systemic and advanced-stage disease when it is diagnosed in more than two-thirds of patients at initial presentation. Follicular lymphoma Grade 1 or 2 with indolent histologic characteristics is presently not considered curable in the majority of patients though it is very sensitive to both chemotherapy and radiotherapy. The policy treated for patients with stage III and IV FL, which recommended by NCCN, is suggested regimens, clinical trial or local RT (palliation) based on the previous results that similar efficacy was obtained after management by chlorambucil single-agent therapy, polychemotherapy, immunochemotherapy, RT or CMT(RT and Chemotherapy). Patients with advanced-stage disease tend to have frequent relapses and the interval between subsequent relapses tends to shorten over time. However, they usually have a relatively long life expectancy, with a median survival ranging from 6 to 10 years. Try to change the natural history of FL and have a long term PFS are the goals of treatment for advanced stage FL.

Since the treatment strategy, watch and wait, was managed in Standford in the 1980s, several prospective randomized trials have failed to demonstrate a survival advantage with immediate treatment versus a "watch and wait" approach in patients with advanced stage, low tumor burden FL. Though many systemic therapy options are available for patients with stage III and IV FL, there is no consensus as to which first-line treatment should be provided to those patients. "Watch and wait" as a approach is still recommended to the patients even in the rituximab era. GELA provided the indications for treatment, when the treatment a patient should be initiated.

The role of traditional RT with or without chemotherapy in advanced stage FL is not definite. FL is considered to be one of the most radiosensitive tumors. However, a significant proportion of patients relapse with systemic disease outside of radiation fields and no difference in OS were observed in advanced patients between RT alone and CMT. The complications related to traditional RT, including cardiovascular disease and disorders of blood cell production, were needed to emphasize for those indolent advanced patients who need frequent palliative management and can long-term survive with NHL. In order to decrease the late complications after Large-field RT, reduction of irradiation field and smaller therapeutic doses of radiation were commonly managed.

Many trials that patients with advanced or recurrent FL managed with very low-dose (4Gy) limited-field RT have shown that high response rates and durable remission can be achieved. The response rates (either a complete or partial response) reported in previous study that low-dose involved-field RT (LD-IFRT) is given in 2 daily fractions (2×2 Gy) is 81% to 92%. The median time to first recurrence was 14 to 15 months. The median overall survival for patients with a positive response was 41 months. The median time to in-field progression was 21months, and the median time to out-field progression was 8 months. The predominant mode of tumor cell death after low-dose RT may be by apoptosis.

Two phase III trials have been designed to assess the further role of LD-IFRT. However, the results have failed to demonstrate the lasting response rate (RR) with LD-IFRT versus in other approaches. The HOVON 47/EORTC 20013 Intergroup study (www.hovon.nl) which compares LD-IFRT to chlorambucil chemotherapy in previously untreated FL patients, the main end points including progression-free survival and quality of life are evaluating. However, the trial was closed in 2005 after 21 cases included because of the clinical adoption of rituximab. The age of most eligible patients was older than 65 years. Another trial, Follicular Radiotherapy Trial (CRUK- FORT), launched recently in the United Kingdom is randomizing patients with FL needing RT to 24 Gy in 12 fractions versus 4 Gy in 2 fractions as either definitive or palliative treatment for FL. A significantly lower overall response rate (81% vs 74%) and 2-year local progression-free rate (94% vs 80%) were found in the 4Gy group. Over half of the patients in the clinic trial were on stage I and stage II. Moreover, the histologies included many other pathologic subtypes of indolent lymphoma besides follicular Grade 1 or 2.

The role of prognostic factors for treatment efficacy is not consensus. Histology has been shown to significantly influence response rates. Compared to other subtypes of indolent lymphoma, the higher response rate of low-dose involved-field radiotherapy (LD-IFRT) as palliative treatment for indolent lymphoma has been explored in follicular lymphoma.

Age at diagnosis, and prior systemic therapy are more estimated. In the retrospective review by Girinsky et al. 48 patients with indolent lymphoma treated with LD-IF-RT, factors that were significantly associated with lack of response including bulky tumor (>5 cm), higher number of prior chemotherapy regimens, and age>65 years. Haas et al. reported their experience of 109 patients with recurrent indolent B-cell NHL treated with LD-IF-RT. Patients with only one or two lymphoma sites and disease size of <5 cm were significantly more likely to achieve a CR.

The management for advanced FL patients with relapse disease after initial management can be affected by significant toxicity associated with Chemotherapy and Radiotherapy. The role of low-dose involved-field radiotherapy (LD-IFRT) as palliative treatment for advanced FL has been explored. LD-IFRT for selected patients including advanced FL, aged lower than 65 years and disease size of <5 cm may have excellent effection in achieving repeated remissions with limited associative toxicity and may postpone the need for systemic therapy. The management is valuable assessed.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female aged range from 18 years to 65 years.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1.
* All patients had histological confirmed follicular lymphoma Grade 1 or 2.
* Recurrent patient with stage III and IV after initial management.
* Had the indications for treatment provided by GELA.
* Rituximab is too expensive to be managed for the patient.
* Adequate organ function.
* Negative pregnancy test.
* Signed informed consent document on file.

Exclusion Criteria:

* Woman who were pregnant or lactating.
* Had uncontrolled metastases in central nervous system.
* With severe local infection or general infective disease.
* Immunotherapy for the treatment of follicular lymphoma within 1 month prior to the start of this trial.
* With other second primary malignancy except cutaneum carcinoma.
* Being or planing to participate in other study.
* Any patient who in the opinion of the investigator should not participate in the study.

Withdrawal Criteria:

* Patient are free to withdrawal completely from the study at any time upon request.
* Patient in the study may be stopped with the patient agreement at any time at the discretion of investigator.
* Continual consolidation chemotherapy after irradiation within the follow-up period.
* In-field progression on irradiation ongoing.
* Poor tolerability adverse events in the period of chemotherapy or irradiation after enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rates - ORR | At day 30 after radiotherapy
Time to treatment failure - TTF | From the start of radiotherapy to the first documented disease progression or death from any cause, whichever occurs first, Assessed up to 40 months.
Number of participants with adverse events with grade 3 or 4 - AEs | The time from the day of treatment to the day of the first documented disease progression or death from any cause, Assessed up to 24 months.
  Toxicity was scored according to the toxicity scale of the National Cancer Institute Common Terminology Criteria for Adverse Events 3.0.

SECONDARY OUTCOMES:
Overall survival - OS | From the initial diagnosis of follicular lymphoma to death from any cause, Assessed up to 100 months.
Rate of in-field progression | From the start of RT to the first documented disease progression within the radiotherapy portal, Assessed up to 24 months.
Rate of out-field progression | From the start of RT to the first documented disease progression outside the radiotherapy field, Assessed up to 40 months.

CONTACTS AND LOCATIONS:
Locations (1):
- DiDeng, Wuhan, Hubei, China